CLINICAL TRIAL: NCT02724735
Title: A Longitudinal Observational Cohort Study of NSI-189, a Neurogenic Compound Among Out-Patients With Major Depressive Disorder
Brief Title: A Longitudinal Observational Cohort Study of NSI-189, With Out-Patients With Major Depressive Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuralstem Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NS2015-2
Record Dates: First submitted 2016-03-15; First posted 2016-03-31 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder (MDD); Major Depressive Disorder; Neurogenesis; Synaptogenesis; NSI-189; Neuralstem
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — NSI-189

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Longitudinal Observational Cohort: Following completion of the NS2014-1 final study visit procedures, Subjects will be offered the opportunity to enroll in this longitudinal observational cohort protocol to monitor their depression and to assess durability of effect and long-term safety of NSI-189.
  Interventions: Drug: NSI-189

INTERVENTIONS:
Drug: NSI-189 — 0 Milligrams, 40 Milligrams or 80 Milligrams administered in the acute study only
  Other Names: NSI-189 Phosphate

SUMMARY:
All subjects completing the randomized treatment period in Protocol NS2014-1 will discontinue study drug and be asked to provide consent to be followed in this 6-month study, at their final safety visit. The study will consist of an enrollment visit, followed by bi-monthly in-clinic visits with monthly telephone visits between in-clinic visits.

DETAILED DESCRIPTION:
Following completion of the NS2014-1 final study visit procedures, Subjects will be offered the opportunity to enroll in this longitudinal observational cohort protocol to monitor their depression and to assess durability of effect and long-term safety of NSI-189.

The Enrollment Visit begins when informed consent is signed.The duration of the follow-up period will be up to 6 months, until the start of a new antidepressant treatment. Subjects who provide consent will be seen for in-person visits every 8 weeks, with bi-monthly phone visits occurring between in-person visits. Safety assessments and efficacy assessments will be performed at each visit. No study drug will be taken during the Longitudinal Observational Cohort study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has the ability to understand the purpose, potential benefits and risks of the study and to provide signed and dated informed consent, authorizing the use of protected health information in accordance with national and local Subject privacy regulations.
2. Subject completed the 12-week randomized treatment period and final study visit for the NS2014-1 clinical study.

Exclusion Criteria:

1. Subjects taking excluded medications.
2. Subject who, in the opinion of the Site Investigator, are unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope and possible consequences of the clinical study.
3. Subject who, in the opinion of the Site Investigator, are unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up and improbability of completing the clinical study.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects having completed the randomized treatment period under the NS2014-1 clinical study protocol.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective: Durability of Effect defined as the time until the start of a new antidepressant treatment (ADT) | 6 months
  The primary objective is to determine the durability of effect of NSI-189 phosphate compared to placebo in subjects with Major Depressive Disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5TH EDITION). Durability of effect is defined as the time until the start of a new antidepressant treatment (ADT).

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 6 months
  Compare the continued Montgomery-Asberg Depression Rating Scale (MADRS) response and remission rates of subjects treated with NSI-189 to those of subjects assigned to placebo. Response is defined as a 50% or greater reduction from baseline to endpoint on the Montgomery-Asberg Depression Rating Scale (MADRS) total score. Remission is defined as an endpoint MADRS total score of 10. The duration of 50% or greater reduction in Montgomery-Asberg Depression Rating Scale (MADRS) total score sustained following treatment will be noted.
Quick Inventory of Depressive Symptomatology - Self-Rated (QIDS-SR) | 6 months
  Compare the continued antidepressant efficacy of NSI-189 with that of placebo.
Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (MGH CPFQ) | 6 months
  Evaluate the continued efficacy of NSI-189 compared to placebo on the cognitive aspects associated with Major Depressive Disorder, and the onset and duration of improvement.
Cogscreen Battery | 6 months
  Evaluate the continued efficacy of NSI-189 compared to placebo on the cognitive aspects associated with Major Depressive Disorder, and the onset and duration of improvement.
Symptoms of Depression Questionnaire (SDQ) | 6 months
  Compare the continued efficacy of NSI-189 with that of placebo, as measured by the Symptoms of Depression Questionnaire (SDQ)
Massachusetts General Hospital Sexual Functioning Inventory (MGH SFI) | 6 months
  Characterize the safety and tolerability of NSI-189, compared to placebo.
The Columbia Suicide Severity Rating Scale (C-SSRS) | 6 months
  Characterize the safety and tolerability of NSI-189, compared to placebo.
17-item Hamilton Depression Rating Scale (HAMD17) | 6 months
  HAMD17 will be used to characterize the safety and tolerability of NSI-189, compared to placebo.
Discontinuation rates | 6 months
  Characterize the safety and tolerability of NSI-189, compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Johe, Ph.D., Study Director — Neuralstem Inc.
Locations (12):
- United States (12):
  - Garden Grove, California
  - National City, California
  - Denver, Colorado
  - Jacksonville, Florida
  - Orlando, Florida
  - Alpharetta, Georgia
  - St Louis, Missouri
  - Staten Island, New York
  - Dayton, Ohio
  - Memphis, Tennessee
  - Dallas, Texas
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Fava M, Johe K, Ereshefsky L, Gertsik LG, English BA, Bilello JA, Thurmond LM, Johnstone J, Dickerson BC, Makris N, Hoeppner BB, Flynn M, Mischoulon D, Kinrys G, Freeman MP. A Phase 1B, randomized, double blind, placebo controlled, multiple-dose escalation study of NSI-189 phosphate, a neurogenic compound, in depressed patients. Mol Psychiatry. 2016 Oct;21(10):1372-80. doi: 10.1038/mp.2015.178. Epub 2015 Dec 8. PMID 26643541